CLINICAL TRIAL: NCT07027020
Title: Efficacy of Intravesical Oxybutynin in Children With Neurogenic Bladder Dysfunction: A Randomized, Prospective Controlled Multi-center Trial
Brief Title: Efficacy of Intravesical Oxybutynin in Children With Neurogenic Bladder Dysfunction
Acronym: POXIPEN
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Farco-Pharma GmbH (Unknown); Ministry of Health, France (Other Government)
Responsible Party: Principal Investigator, LEMELLE Jean-Louis, Principal investigator, head of paediatric surgery, Central Hospital, Nancy, France
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019PI119; 2022-501902-36-00 (EU CTIS Number)
Record Dates: First submitted 2025-05-22; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Spina Bifida
Keywords: Intravesical Oxybutynin; overactive neurogenic bladder; intermittent catheterization; Oxybutynin; anticholinergic; Pediatric patients
MeSH Terms: conditions — Spinal Dysraphism | interventions — oxybutynin; Administration, Intravesical

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- IntraVesical Oxybutynin (IVO) (Experimental): Instillation of oxybutynin conditioned in VESOXX® 10mg/10mL ready-to-use syringes (1mg/mL) at the end of the evacuation catheterization.
  Dose: 0.4mg/kg/day in 2 to 3 instillations per day, i.e. a maximum of 10mg per instillation. Maximum dose: 20mg/day for patients aged 6-11 years and 11 months, and 30mg/day for patients aged 12-17 years.
  Interventions: Drug: Oxybutynin Hydrochloride
- IntraVesical Placebo (PCB) (Placebo Comparator): Instillation of saline solution conditioned in 10 mL ready-to-use syringes at the end of the evacuation catheterization. Dose equivalent to IVO in ml, i.e. always 0.4mg/kg/day, i.e. a maximum of 10 mL per instillation. Maximum dose: 20mL/day for patients aged 6-11 years and 11 months, and 30mL/day for patients aged 12 to 17 years.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxybutynin Hydrochloride — Pharmaceutical form: solution. Route of administration: Intravesical. Medicinal product unique ID: PRD8074745. EU active substance code: SUB03581MIG.
  Arms: IntraVesical Oxybutynin (IVO)
Drug: Placebo — Pharmaceutical form: solution. Route of administration: Intravesical.
  Other Names: Sterile 0.9% NaCl solution for intravesical instillation
  Arms: IntraVesical Placebo (PCB)

SUMMARY:
Malformation of the lumbosacral region (spina bifida) affects the innervation of the bladder in children. The usual evolution leads to a neurological bladder with small capacity, poor compliancy and overactivity, exposing to incontinence and obstruction to the evacuation of urine. It is responsible for renal failure requiring dialysis and transplantation. Current therapeutics aim to evacuate urine and reduce intravesical pressure. It gradually combines 1) intermittent catheterization, 2) anticholinergics, 3) botulinum toxin (Botox®) injection into the detrusor (bladder muscle) by cystoscopy and 4) surgery (vesicostomy, Bricker, enterocystoplasty). Oxybutynin relaxes the detrusor, improves continence and reduces intravesical pressure. It is usually administered per os, but there are contraindications (glaucoma, myasthenia), side effects (constipation, dry mouth). It can be difficult to swallow for children, and drug resistance may develop. It can lead to ineffective treatment requiring therapeutic escalation. The next step, intradetrusor Botox® injection, is invasive (cystoscopy), has a limited duration of action (6 months) and must be performed under general anesthesia in children.

Surgical treatments are effective but irreversible and responsible for morbidity and mortality. A randomized study was performed demonstrating the efficacy of intravesical oxybutynin compared to oral administration in adult patients. This study found a significant increase in bladder capacity and a significant decrease in side effects in the intravesical oxybutynin group. Due to the relative difficulties of intravesical oxybutynin delivery (preparation, cost) and the more invasive nature, it is not used as an alternative to oral oxybutynin.

Our hypothesis is that this treatment may have a legitimate place in the treatment of neurogenic bladder in patients with failure of anticholinergic treatment before a therapeutic escalation requiring an invasive procedure (Botox®, enterocystoplasty) especially in children for whom repeated general anesthesia for Botox® injection may interfere with brain development. In this way, we aim to extend the time to therapeutic escalation in the pediatric population.

The main objective of the trial is to compare the efficacy on maximal bladder capacity of intravesical oxybutynin instillation versus placebo in the treatment of children with overactive neurogenic bladder (spina bifida), performing intermittent catheterization, for whom oral anticholinergic treatment is ineffective or poorly tolerated.

DETAILED DESCRIPTION:
Secondary objectives of the trial :

* Secondary efficacy objectives will be analyzed following a fixed sequence in a priori ordered hypotheses: to evaluate after treatment with intravesical oxybutynin (IVO) or placebo instillation: maximum bladder pressure evolution; incontinence: time to clinical treatment failure perceived by the patient. These parameters are considered by experts to be objective markers of neurological bladder improvement, in addition to the primary urodynamic objective.
* Evaluate and compare between groups the tolerance and adverse effects of treatment.
* Evaluate and compare between groups the number of responders and continent patients after treatment
* Evaluate and compare between groups the usability of Intravesical Oxybutynin.
* Evaluate and compare between groups the evolution of quality of life.
* Evaluate and compare between groups the evolution of bladder diary data.
* Evaluate and compare between groups the evolution of other urodynamic parameters.
* Evaluate and compare between groups the evolution of renal ultrasonography parameters.
* Identify factors, among the patient's characteristics, associated with a greater probability to be a responder or non-responder to intravesical oxybutynin.

ELIGIBILITY:
Inclusion Criteria:

* Person affiliated to or beneficiary of a social security plan
* In failure of treatment with one or more anticholinergics defined by a response considered insufficient by the investigator after at least 4 weeks of optimal dose treatment, unable to take oral oxybutynin or intolerable adverse events
* Having performed renal ultrasonography less than 2 months ago
* Having performed cystomanometry less than 6 months ago including maximal bladder capacity and maximal bladder pressure (preferably not under oral oxybutynin treatment)
* Age between 6 and 17 years old
* Informed about study organization, having given consent to participate and each legal representative have signed the informed consent
* Having undergone the medical examination adapted to research
* Presenting overactive bladder due to spina bifida confirmed by urodynamic check-up of less than 6 months. Overactive bladder is defined according to International Children's Continence Society, (ICCS): "a urodynamic observation characterized by involuntary detrusor contractions during the filling phase which may be spontaneous or provoked"
* Carrying out intermittent catheterization for at least 6 weeks and at least three times a day
* Able and volunteer to perform intravesical catheterization and instillation (patient or parents).

Exclusion Criteria:

* Person displaying known allergy to one of the components of evaluated product (notably oxybutynin).
* Person with congestive cardiac failure
* Person with cardiac arrhythmia
* Person with tachycardia
* Person with uncontrolled hypertension
* Person under one of the following treatments : Bisphosphonates; Cytochrome P450 Inhibitors (such as ketoconazole and Erythromycin); Cholinesterase inhibitors.
* Person displaying a contraindication to evaluated product, in particular: Hypersensitivity to oxybutynin; Myasthenia; Angle-closure glaucoma; Functional or organic gastrointestinal obstruction including pyloric stenosis, paralytic ileus and intestinal atony; Serious gastro-intestinal disorders (e.g., severe ulcerative colitis and toxic megacolon); Patients who have undergone ileostomy, colostomy, severe hemorrhagic colectasis or rectocolitis; Subvesical obstruction (urethral stenosis, posterior urethra valve); Ongoing treatment with anticholinergic drugs for another indication that could not be stopped; Patient with polyuria of other origin (renal, heart, potomania); Concomitant oxygenotherapy.
* Woman of childbearing age without highly effective contraception (Sexual abstinence OR combined contraception by oral, intravaginal or transdermal ovulation inhibition OR progestin-only contraception by oral, injectable or implantable ovulation inhibition OR Intrauterine device or hormonal IUD).
* Pregnant, parturient or breastfeeding woman.
* Person deprived of liberty for judicial or administrative decision.
* Person under psychiatric care as referred in articles L. 3212-1 and L. 3213-1.
* Intradetrusor injection of botulinum toxin less than 6 months before.
* Person with hyperthyroidism
* Person with coronary cardiac disease.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Evolution of maximal bladder capacity at 4 weeks of treatment (end of follow-up) | 4 weeks
  This parameter is considered by experts to be an objective marker of improvement in neurological bladder, in addition to the secondary clinical objective. It was used as the primary objective in the only prospective study in the literature.
  It is obtained by cystomanometry and is defined by the maximum volume (in mL) measured at the moment when permission to urinate is given to the patient, after filling via urethral catheter. In younger patients, urination occurs spontaneously, and this value is obtained a posteriori by curve analysis.
  If treatment is successful, maximum bladder capacity should increase.

SECONDARY OUTCOMES:
Evolution of maximal bladder pressure at 4 weeks of treatment (end of follow-up) | 4 weeks
  This parameter is considered by experts to be an objective marker of neurological bladder improvement, in addition to the primary objective.
  This data is obtained during cystomanometry. If treatment is effective, it should decrease.
Urinary incontinence | 4 weeks
  Time to clinical treatment failure defined by criteria found in literature and marketing authorization of Botox® in a 28-day time frame (at least one of the 3 criteria):
  * Treatment judged as non-effective by either the patient or the practitioner;
  * Reduction of urinary incontinence to less than 50% of the initial occurrences measured in the initial bladder diary;
  * Intolerable side effects reported by the patient.
Evaluation of the number of side effects | 4 weeks
  Side effects are recorded by the patient in a treatment follow-up booklet or by the practitioner during follow-up. They include digestive, psychiatric, neurological, cutaneous and urological disorders, pain associated with instillation of the product, and other effects.
Proportion of responders at 4 weeks of treatment | 4 weeks
  This corresponds to patients who achieved at least a 50% reduction in urinary incontinence episodes after 4 weeks of treatment, with no intolerable side effects (leading to discontinuation of treatment) at the end of the study. The number of incontinence episodes are collected over 72 consecutive hours in the week preceding each visit (V1, V2 and V3) by the patient on a bladder diary. Side effects are recorded by the patient in the treatment follow-up booklet and by the practitioner at each visit.
Proportion of continent patients at 4 weeks of treatment | 4 weeks
  It corresponds to patients who had a 100% reduction in urinary incontinence episodes by the end of the study. This group is part of the responder group at 4 weeks of treatment.
Product usability measured with usability questionnaire | 4 weeks
  Ease of use, which improves patient acceptability and compliance, is measured using the short version of the Usability Metric for User Experience scale (UMUX-LITE) containing two positive items with a 7-point response scale, coupled with six ad hoc questions specific to the treatment and the disease. The values of each question range from 0 (totally disagree) to 7 (totally agree).
Standardized difference in patient quality of life calculated according to the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF) score between the beginning and the end of the study. | 4 weeks
  It is calculated on the basis of changes in the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF) questionnaire score between the start and end of the patient's participation in the study. The answers to the 3 items of the questionnaire result in a sum, with minimum score of 0 ("no incontinence"), and maximum score of 21 ("maximum urinary incontinence").
Standardized difference in patient quality of life calculated according to the KIDSCREEN-10 score between the beginning and the end of the study. | 4 weeks
  It is calculated on the basis of changes in the KIDSCREEN-10 Index between the start and end of the patient's participation in the study. The KIDSCREEN-10 Index, developed by the project "Screening For and Promotion of Health-Related Quality of Life in Children and Adolescents - a European Public Health perspective", contains 10 items. The sum score is comprised between 10 and 50, where 10 represents the lowest possible value and thus a very low health-related quality of life and 50 the maximum value, i.e. a very high health-related quality of life.
Evolution of the number of urinary catheterizations at 4 weeks of treatment | 4 weeks
  This evolution is assessed by comparing the number of urinary catheterizations over 72 hours during the week preceding each visit (V1, V2 and V3).
Evolution of the volume of urinary catheterizations at 4 weeks of treatment | 4 weeks
  This evolution is assessed by comparing the volume of urinary catheterizations over 72 hours during the week preceding each visit (V1, V2 and V3).
Evolution of the bladder compliance at 4 weeks of treatment | 4 weeks
  The bladder compliance (mL/cmH2O) is measured 2 times using cystomanometry : prior to treatment and at the end of treatment. The 2 values obtained are compared.
Evolution of the minimum filling volume causing uninhibited detrusor contraction at 4 weeks of treatment | 4 weeks
  The minimum filling volume causing uninhibited detrusor contraction (mL) is measured 2 times using cystomanometry : prior to treatment and at the end of treatment. The 2 values obtained are compared.
Evolution of the Detrusor leak point pressure at 4 weeks of treatment | 4 weeks
  The Detrusor leak point pressure (cmH2O) is measured 2 times using cystomanometry : prior to treatment and at the end of treatment. The 2 values obtained are compared.
Evolution of the volume of bladder filling during urine loss at 4 weeks of treatment | 4 weeks
  The volume of bladder filling during urine loss (mL) is measured 2 times using cystomanometry : prior to treatment and at the end of treatment. The 2 values obtained are compared.
Evolution of renal ultrasonography at 4 weeks of treatment | 4 weeks
  Renal ultrasonography performed at the end of treatment is compared with the renal ultrasonography performed prior to treatment. This enables an assessment of the impact on the upper urinary tract, and is an indirect marker of bladder condition. The standard parameters assessed are :
  * Anteroposterior diameter of the pyelo (mm);
  * Ureter diameter (mm)

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire De Bordeaux, Bordeaux
  - Centre Hospitalier Régional Et Universitaire De Brest, Brest
  - Centre Hospitalier Universitaire De Caen Normandie, Caen
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Centre Hospitalier De Colmar, Colmar
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - Centre Hospitalier Universitaire de Lille, Lille
  - Centre Hospitalier Et Universitaire De Limoges, Limoges
  - Centre Hospitalier Régional De Marseille, Marseille
  - Fondation Lenval Nice, Nice
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Trousseau (chirurgie viscérale pédiatrique et néonatale), Paris
  - Hôpital Trousseau (médecine physique et de réadaptation pédiatrique), Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Hospitalier Universitaire De Saint Etienne, Saint-Etienne
  - Les Hopitaux Universitaires De Strasbourg, Strasbourg
  - Centre Hospitalier Régional Et Universitaire de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buzzi M, Epstein J, Hatem Z, Juge N, Mazeaud C, Lemelle JL, Berte N. Intravesical oxybutynin for bladder capacity in children with spina bifida: the 'Place de l'OXybutynine Intravesicale chez le Patient Enfant Neurologique' (POXIPEN) trial protocol. BJU Int. 2026 Feb;137(2):390-398. doi: 10.1111/bju.70058. Epub 2025 Nov 3. PMID 41178302
- See also: Clinical Trials — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2022-501902-36-00